CLINICAL TRIAL: NCT01344278
Title: Comparative Effectiveness of Diabetes Prevention Strategies in Women With GDM
Brief Title: Diabetes Prevention Strategies in Women With Gestational Diabetes Mellitus (GDM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01HS019367-01 (AHRQ)
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Gestational Diabetes; Obesity
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Counseling (Experimental)
  Interventions: Behavioral: Lifestyle Counseling
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle Counseling — A lifestyle curriculum of individualized telephone counseling calls, augmented with e-mails and an interactive study Web site.
  Arms: Lifestyle Counseling

SUMMARY:
The main goal of this study is to examine the comparative effectiveness of diabetes prevention strategies in women with Gestational Diabetes Mellitus (GDM) on the control of the following conditions: obesity, hyperglycemia, hypertension and depression. This randomized lifestyle intervention study will be conducted at Kaiser Permanente Northern California. Women in the intervention will receive a letter on gestational weight gain during pregnancy and in the postpartum period, a curriculum of individualized lifestyle counseling via telephone, augmented with e-mail and an interactive Web site. Patients randomized to the usual care arm will receive the standard-care telephone calls from the Perinatal Center during pregnancy and the Center's printed educational materials postpartum. Outcomes will be assessed through the electronic medical record and patient surveys conducted during pregnancy and at 6-weeks, 6- months and 1-year postpartum.

ELIGIBILITY:
Inclusion Criteria:

All women, 18 years of age or older, receiving medical care at Kaiser Permanente Northern California with a pregnancy complicated by gestational diabetes between March 2011 and May 2012 that have a telephone or cellular phone will be eligible.

Exclusion Criteria:

Women with overt diabetes not recognized prior to pregnancy (any women with fasting plasma glucose > 126 mg/dl, or any plasma glucose level over 200 mg/dl on more than 1 occasion during pregnancy) will be excluded from the analyses but will be eligible for the lifestyle intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2480 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome: meeting the postpartum weight goal | through 12 months postpartum
  Will be the proportion of women who reach their postpartum weight goal (based on their pre-pregnancy weight) and the total amount of weight change (in kilograms).
  Weight goals:
  a) reaching pre-pregnancy weight if women had a normal pre-pregnancy weight; or b) achieving a 5% reduction from pre-pregnancy weight if overweight or obese prior to pregnancy.

SECONDARY OUTCOMES:
Blood pressure | through 12 months postpartum
Depression | through 12 months postpartum
Glycemia | through 12 months postpartum
percent of calories from fat | through 12 months postpartum
physical activity | through 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Assiamira Ferrara, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Division of Research Northern California, Oakland, California, United States

REFERENCES:
- [Derived] Gadgil MD, Ehrlich SF, Zhu Y, Brown SD, Hedderson MM, Crites Y, Ferrara A. Dietary Quality and Glycemic Control Among Women with Gestational Diabetes Mellitus. J Womens Health (Larchmt). 2019 Feb;28(2):178-184. doi: 10.1089/jwh.2017.6788. Epub 2018 Oct 30. PMID 30376391
- [Derived] Hedderson MM, Brown SD, Ehrlich SF, Tsai AL, Zhu Y, Quesenberry CP, Crites Y, Ferrara A. A Tailored Letter Based on Electronic Health Record Data Improves Gestational Weight Gain Among Women With Gestational Diabetes Mellitus: The Gestational Diabetes' Effects on Moms (GEM) Cluster-Randomized Controlled Trial. Diabetes Care. 2018 Jul;41(7):1370-1377. doi: 10.2337/dc17-1133. Epub 2018 Apr 18. PMID 29669736
- [Derived] Ferrara A, Hedderson MM, Brown SD, Albright CL, Ehrlich SF, Tsai AL, Caan BJ, Sternfeld B, Gordon NP, Schmittdiel JA, Gunderson EP, Mevi AA, Herman WH, Ching J, Crites Y, Quesenberry CP Jr. The Comparative Effectiveness of Diabetes Prevention Strategies to Reduce Postpartum Weight Retention in Women With Gestational Diabetes Mellitus: The Gestational Diabetes' Effects on Moms (GEM) Cluster Randomized Controlled Trial. Diabetes Care. 2016 Jan;39(1):65-74. doi: 10.2337/dc15-1254. Epub 2015 Dec 9. PMID 26657945
- [Derived] Ferrara A, Hedderson MM, Albright CL, Brown SD, Ehrlich SF, Caan BJ, Sternfeld B, Gordon NP, Schmittdiel JA, Gunderson EP, Mevi AA, Tsai AL, Ching J, Crites Y, Quesenberry CP Jr. A pragmatic cluster randomized clinical trial of diabetes prevention strategies for women with gestational diabetes: design and rationale of the Gestational Diabetes' Effects on Moms (GEM) study. BMC Pregnancy Childbirth. 2014 Jan 15;14:21. doi: 10.1186/1471-2393-14-21. PMID 24423410
- See also: GEM Trial Publication — http://www.ncbi.nlm.nih.gov/pubmed/26657945